CLINICAL TRIAL: NCT02200224
Title: Clinical Utility of Rapid CT/NG Testing in the ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Rich Rothman, Professor, Vice Chair of Research, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: JHUIRB00026782; U54EB007958 (NIH)
Record Dates: First submitted 2014-07-23; First posted 2014-07-25 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Sexually Transmitted Diseases
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rapid Testing/Treatment Group (Experimental): All subjects enrolled in the rapid testing group will receive rapid CT/NG and TV testing in addition to the CT/NG Nucleic Acid Amplification Test (NAAT) and wet mount testing that is currently used in the ED.
  Interventions: Other: Rapid Testing
- Control (No Intervention): All subjects enrolled in the control group will receive CT/NG and TV testing according to the current standard of care for Johns Hopkins ED.

INTERVENTIONS:
Other: Rapid Testing
  Arms: Rapid Testing/Treatment Group

SUMMARY:
The purpose of this study is to:

1. determine the clinical impact of rapid Chlamydia Trachomatis (CT), Neisseria Gonorrhoeae (NG) testing on antibiotic over and under treatment for CT/NG in women evaluated in the Emergency Department (ED) for a Sexually Transmitted Infection (STI).
2. determine the clinical impact of rapid Trichomonas Vaginalis (TV) testing on antibiotic under and over treatment for TV in women evaluated in the ED for an STI
3. evaluate the feasibility of integrating rapid Chlamydia Trachomatis (CT), Neisseria Gonorrhoeae (NG) and TV testing in the Emergency Department setting.

To evaluate the impact or rapid CT/NG/TV testing an patient comprehension of Sexually Transmitted Infection diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* The study population includes women between the age of 18 and 50 who present to the ED and are going to receive CT/NG testing in the ED.

Exclusion Criteria:

* Patients will be excluded if they are unable to provide informed consent or are not English speaking.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Overtreatment rate of CT/NG between the control and interventional groups | 2 week follow-up
  Overtreatment is defined as CT/NG negative patients who received antibiotic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Dugas, MD,PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaydos CA, Ako MC, Lewis M, Hsieh YH, Rothman RE, Dugas AF. Use of a Rapid Diagnostic for Chlamydia trachomatis and Neisseria gonorrhoeae for Women in the Emergency Department Can Improve Clinical Management: Report of a Randomized Clinical Trial. Ann Emerg Med. 2019 Jul;74(1):36-44. doi: 10.1016/j.annemergmed.2018.09.012. Epub 2018 Nov 2. PMID 30392736